CLINICAL TRIAL: NCT02161432
Title: Relative Bioavailability of a BI 187004 Tablet Formulation in Comparison With an Oral Solution and the Influence of Food on the Bioavailability of the Tablet Formulation (a Randomised, Open-label, Single Dose, Three-way Crossover Trial in Healthy Subjects)
Brief Title: Relative Bioavailability of a BI 187004 Tablet Formulation in Comparison With an Oral Solution and the Influence of Food on the Tablet Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1307.3; 2013-004627-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Healthy

ARMS (3):
- Treatment A (Experimental): single dose of BI 187004 in fasted state
  Interventions: Drug: BI 187004
- Treatment B (Experimental): single dose of BI 187004
  Interventions: Drug: BI 187004
- Treatment C (Experimental): single dose of BI 187004 in fed state
  Interventions: Drug: BI 187004

INTERVENTIONS:
Drug: BI 187004 — single dose BI 187004 given as tablet in fed state
  Arms: Treatment C
Drug: BI 187004 — single dose BI 187004 given as tablet in fasted state
  Arms: Treatment A
Drug: BI 187004 — single dose BI 187004 given as oral solution
  Arms: Treatment B

SUMMARY:
To determine the relative bioavailability of an BI 187004 tablet formulation compared to an oral solution of BI 187004 and to assess the influence of food on the bioavailability of the tablet formulation.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. Age of 18 to 50 years
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2

Exclusion criteria:

1. Any finding in the medical examination (including BP, pulse rate (PR) or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) of BI 187004 | up to 17 days postdose
Cmax (maximum measured concentration of the analyte in plasma) of BI 187004 | up to 17 days postdose

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 17 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1307.3.1 Boehringer Ingelheim Investigational Site, Biberach, Germany